CLINICAL TRIAL: NCT06968507
Title: Comparison of the Effectiveness of Oral and Intratympanic Corticosteroid Treatments in Patients Diagnosed With Sudden Sensorineural Hearing Loss
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Koray Islek, Resident Doctor, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: kartalentdepartment
Record Dates: First submitted 2025-04-21; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Sudden Sensorineural Hearing Loss
Keywords: intratympanic dexamethasone; Sudden sensorineural hearing loss; oral methylprednisolone
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Methylprednisolone; Pharmaceutical Preparations; Dexamethasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oral methylprednisolone treatment (Active Comparator): Group 1 included patients who received oral methylprednisolone treatment daily for 2 weeks (48 mg for the first 7 days, 32 mg for the following 2 days, 16 mg for the 2 days, and 8 mg for the last 3 days).
  Interventions: Drug: Methylprednisolone (drug)
- intratympanic dexamethasone treatment (Active Comparator): Group 2 included patients who received intratympanic 8 mg/2 ml dexamethasone every other day, totally 4 doses.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Methylprednisolone (drug) — In our study, we use methylprednisolone as a oral treatment daily for 2 weeks (48 mg for the first 7 days, 32 mg for the following 2 days, 16 mg for the 2 days, and 8 mg for the last 3 days)
  Arms: oral methylprednisolone treatment
Drug: Dexamethasone — In our study we use dexamethasone 8mg/2ml form as intratympanic treatment every other day, totally 4 doses.
  Arms: intratympanic dexamethasone treatment

SUMMARY:
The goal of this clinical trial is to learn which one works to treat better in patients with sudden sensorineural hearing loss, oral or intratympanic corticosteroid treatment.

The main question it aims to answer is:

Which corticosteroid treatment is more effective in patients with sudden sensorineural hearing loss, oral or intratympanic?

* In our study, it was planned to divide the treatment schemes compared into two groups. Group 1 included patients who received oral methylprednisolone treatment daily for 2 weeks (48 mg for the first 7 days, 32 mg for the following 2 days, 16 mg for the 2 days, and 8 mg for the last 3 days). Group 2 included patients who received intratympanic 8 mg/2 ml dexamethasone every other day, totally 4 doses.
* Visit the clinic after diagnose in first week, second week, first month and second month for checkups and tests ( temporal MR, odimetric results)

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Unilateral sudden sensorineural hearing loss that developed within 72 hours and has lasted for 14 days or less
* Affected side PTA (500-100-2000-4000hz) should be over 50dB
* Affected side should be at least 30dB lower than healthy side in 3 frequencies
* Hearing should be symmetrical according to patient's statement before sensorineural hearing loss
* If used, steroid use should be less than 10 days
* Cerebellar and vestibular examination should be normal

Exclusion Criteria:

* Having a history of hearing-related surgery other than a ventilation tube
* Having a history of previous hearing loss, fluctuating hearing or Meniere's disease, chronic inflammatory or suppurative ear disease or cholesteatoma, otosclerosis
* Being under 18 or over 80
* Having a history of physical-barotrauma
* Presence of structural or retrocochlear pathology in the examination and imaging that would explain the unilateral hearing loss
* Patients diagnosed with tuberculosis or receiving prophylactic tuberculosis treatment, diabetes mellitus, rheumatological patients, those with atherosclerotic disease, serious psychiatric patients, those receiving chemotherapy, radiotherapy or immunosuppressant treatment, pancreatitis patients, HIV, hepatitis C and B patients, those with chronic renal failure, substance abusers, those with active herpetic lesions, severe osteoporosis patients, those with hearing loss within 4 weeks after general anesthesia, those with a history of head and neck cancer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2028-09-10 (Estimated); Study Completion 2028-09-10 (Estimated)

PRIMARY OUTCOMES:
odiometric hearing results (PTA) | from the begining of the treatment in first, second week and first second month
  Pure tone audiometry yields hearing threshold values and speech audiometry yields a word recognition score, the highest percentage (0%-100%; normal >90%) of monosyllabic words identified correctly from digitally recorded standardized 50-word lists presented to each ear of each participant. The primary end point of the study was the change in hearing threshold (dB PTA) from the first audiogram to the 2-month follow-up audiogram. We will define intratympanic or oral treatment to be inferior to other one if the mean post-treatment change in dB PTA of the oral group or intratympanic group exceeds that of the other one by more than 10 dB. Our standard audiometric measure (10 dB) is widely considered the smallest change boundary for clinical reporting of asymetries and air-bone gaps for clinical test procedures (Dirks D. Factors related to bone conduction reliability. Arch Otolaryngol. 1964;79:551-558.)

CONTACTS AND LOCATIONS:
Overall Officials: Rasim Yılmazer, Study Director — Dr. Lutfi Kirdar Kartal Training and Research Hospital
Locations (1):
- Dr Lütfi Kırdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- See also: Oral vs intratympanic corticosteroid therapy for idiopathic sudden sensorineural hearing loss: a randomized trial — https://pubmed.ncbi.nlm.nih.gov/21610239/
- See also: FACTORS RELATED TO BONE CONDUCTION RELIABILITY — https://pubmed.ncbi.nlm.nih.gov/14135072/